CLINICAL TRIAL: NCT02302820
Title: Nurse-led Patient-centered Advance Care Planning: A Pilot Study
Acronym: ACP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Diane Holland, Clinical Nurse Researcher, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 14-006947
Record Dates: First submitted 2014-10-03; First posted 2014-11-27 (Estimated); Last update posted 2016-01-05 (Estimated); Status verified 2016-01

CONDITIONS: Advance Care Planning; Nurse Care Coordination; Multiple Chronic Health Conditions
Keywords: Advance Care Planning; Nurse Care Coordination; Comparative Effectiveness; Advance Directive; Decision Aides
MeSH Terms: conditions — Multiple Chronic Conditions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Make Your Wishes Known (Active Comparator): A Decision Aid that uses interactions, videos, vignettes.
  A formatted Advance Directive; saved data that may be revisited to produce a revised Advance Directive
  Interventions: Other: Advance Care Planning Intervention
- Mayo Clinic-Advance Health Care Planning (Active Comparator): Not an online decision aid
  Written instructions, worksheets, and Advance Directive to complete
  Interventions: Other: Advance Care Planning Intervention
- Mydirectives.com (Active Comparator): Online decision aid that uses interactions, videos, and vignettes.
  An electronically stored Advance Directive that may be printed.
  Interventions: Other: Advance Care Planning Intervention
- Prepare (Active Comparator): An online decision aid that uses interactions, videos and vignettes.
  A printed summary useful for transposing values and treatment wishes into an Advance Directive; a list of action steps.
  Interventions: Other: Advance Care Planning Intervention

INTERVENTIONS:
Other: Advance Care Planning Intervention — ACP Intervention The ACP intervention involves structured discussions between patients and NCCs using 1 of 4 decision aids in order to clarify patient's values, goals and preferences for "living well" and sharing goals with family, SDM/HCA, and the health care team. Because the time needed for reflective thinking, decision making and discussions with family are important components of the ACP process, the intervention is designed to occur in at least 3 NCC/patient visits over approximately 4 weeks. The NCC will assist patients in the ACP process following scripts specific to each of the decision aids.

SUMMARY:
This study begins to look at ways nurses in primary care might help patients engage in Advance Care Planning and communicate their values and preferences to family and doctors.

DETAILED DESCRIPTION:
The purpose of this pilot study is to determine the feasibility and acceptability of study procedures in comparing the effectiveness of four advance care planning (ACP) decision aids when used by Nurse Care Coordinators (NCCs) with their patients in primary care. Study activities include face-to-face participation in primarily 3 one-hour meetings with their NCC and completion of study questionnaires at baseline and at completion of the intervention. If during the ACP process the patient identifies a surrogate decision maker/health care agent (SDM/HCA), the SDM/HCA will be invited to also participate in the study by answering a questionnaire when the patient has completed the ACP intervention.

Findings from prior studies provide evidence of the success of the ACP decision aids for use in the ACP process. The proposed study is a logical next step to meet the need to enhance patient-centeredness in primary care practices. The study team is strategically positioned to successfully conduct the proposed study with adequate support and skills available. The proposed study is innovative in that it compares the effectiveness of evidence-based ACP decision aids when used by primary care nurses in collaboration with the patients they serve.

A four-arm, prospective, comparative, feasibility design is proposed. Participants will be recruited from the caseloads of NCCs from Mayo Clinic's primary care practice. After enrollment patients will be randomly assigned to either one of 3 ACP web-based decision aids or an ACP educational brochure decision aid arm to receive education and guidance related to the ACP process.

The central hypothesis is that ACP by NCCs in collaboration with patients in primary care settings is feasible and effective when supported by a decision aid. All 4 ACP decision aids have been proven successful when used by patients independently, but no evidence exists regarding their success when used in a patient/clinician collaboration in primary care. Group differences will direct us to explore whether one or more ACP decision aid performs better than others, thereby indicating that successful ACP by NCCs in primary care settings may be supported by particular decision aids. Direct benefits to subjects involved are not assured, but information regarding the ACP process and the possibility of identifying a surrogate decision maker and completion of an advance directive provides a potential benefit.

ELIGIBILITY:
Patients on the list of each NCC who do not have an Advance Directive on file in the Mayo electronic health record will be invited to participate.

Inclusion Criteria: This study will include community-dwelling adult patients with multiple chronic health conditions who do not have an Advance Directive document on file and their SDM/HCA if identified during the course of the intervention. We will accrue 40 patients and up to 40 SDM/HCAs to participate in this pilot study as subjects (80 total participants).

Exclusion Criteria: Because the ACP process, as part of self-management, is a deliberative process, patients with dementia or a serious, persisting psychiatric diagnosis identified in the medical record will be excluded. Patients whose cannot speak or read English will be excluded since it is beyond the scope of this pilot study to employ interpreters.

No vulnerable populations will be included in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2014-12; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Composite Measure of Acceptability and Feasibility | 4 months
  Data regarding acceptability and feasibility of the study methods will be recorded following CONSORT Guidelines to monitor accrual and retention and include the percent of patients eligible for the study over the study period; percent of patients who are approached and accept study participation, percent of patients who complete the intervention and percent of forms completed. Patient satisfaction with the ACP decision aids will be measured using the Patient Satisfaction with ACP Survey.

SECONDARY OUTCOMES:
Composite Measure of Effects and Comparisons of the Four ACP Decision Aids | 4 months
  To conduct preliminary effects and comparisons of the four ACP decision aids, the ACP Engagement Survey consisting of Process and Action components will be mailed to the patient or administered via a telephone call by the study coordinator after the intervention is completed. There are 31 Process questions organized into 4 subscales, each with a Likert response set ranging from 1-5. There are 19 dichotomous (yes/no) Action measure questions. The formal identification of a SDM/HCA and the proportions of Advance Directives will be obtained from patients' electronic health records. Names of SDM/HCAs and Advance Directive documents are stored in a specific location with the electronic health record. The study coordinator will review the electronic health record for SDM/HCA and an advance directive one month after the patient has completed the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Diane Holland, RN, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States